CLINICAL TRIAL: NCT00042484
Title: Community Organizing Network for Environmental Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Other Study IDs: 10688-CP-001
Record Dates: First submitted 2002-07-30; First posted 2002-08-01 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Asthma
Keywords: Asthma; Children's Health; Community Based Research
MeSH Terms: conditions — Asthma

INTERVENTIONS:
Procedure: Community-level intervention & policy change

SUMMARY:
The Community Organizing Network for Environmental Health is a part of Community Action Against Asthma (CAAA), which, in turn is a part of the Michigan Center for the Environment and Children's Health. It is a community-based intervention research partnership between the University of Michigan, community-based organizations, and health care institutions in Detroit.

DETAILED DESCRIPTION:
The aims of the Community Organizing Network for Environmental Health are to:

* share with community groups and organizations the findings from data collected through household and air quality research of the CAAA project;
* identify and engage existing community groups and organizations interested in working on environmental issues important to their neighborhood and community in the hopes of creating an interorganizational network (I.N.);
* work with member group of the I.N. to organize, coordinate and conduct activities to reduce physical environmental threats related to asthma; and
* increase community awareness and knowledge of factors associated with the environment and asthma through sharing of findings to community residents through presentations, annual reports, postings of websites, and community forums

Age Groups: Child, Adult, Older Adult
Dates: Primary Completion 2002-06 (Actual); Study Completion 2002-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan School of Public Health, Ann Arbor, Michigan, United States